CLINICAL TRIAL: NCT02109198
Title: Cranial-nerve Non-invasive Neuromodulation (CN-NINM) for Balance Deficits After Mild Traumatic Brain Injury (Pilot Phase)
Brief Title: Cranial-nerve Non-invasive Neuromodulation (CN-NINM) for Balance Deficits After Mild Traumatic Brain Injury (Pilot Trial)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: protocol withdrawn
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Virginia Commonwealth University (Other); US Department of Veterans Affairs (U.S. Federal Agency); The Defense and Veterans Brain Injury Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CN-NINM pilot
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active CN-NINM PoNS (Experimental): Active CN-NINM PoNS - Active cranial-nerve non-invasive neuromodulation (CN-NINM) using the Portable Neuromodulation Stimulator (PoNS) and balance/gait rehabilitation with physical therapy
  Interventions: Device: Active CN-NINM PoNS
- Sham PoNS CN-NINM (Placebo Comparator): Sham CN-NINM PoNS - Sham cranial-nerve non-invasive neuromodulation (CN-NINM) using the Portable Neuromodulation Stimulator (PoNS) and balance/gait rehabilitation with physical therapy
  Interventions: Device: Sham CN-NINM PoNS

INTERVENTIONS:
Device: Active CN-NINM PoNS — Delivery of active stimulation of the tongue during in-person therapy sessions (1 hour) and during two home sessions (40 minutes) daily on 6 of 7 days per week (120 total sessions). Stimulation sessions will be separated by at least 4 hours.
  Other Names: Active cranial-nerve non-invasive neuromodulation (CN-NINM); Portable Neuromodulation Stimulator (PoNS)
  Arms: Active CN-NINM PoNS
Device: Sham CN-NINM PoNS — Delivery of sham stimulation of the tongue during in-person therapy sessions (1 hour) and during two home sessions (40 minutes) daily on 6 of 7 days per week (120 total sessions). Stimulation sessions will be separated by at least 4 hours.
  Arms: Sham PoNS CN-NINM

SUMMARY:
The purpose of this study is to determine the feasibility of combining PoNS therapy with standard vestibular and balance therapy with the proposed double-blind design; evaluate preliminary indications of efficacy. This study is also evaluating recruitment rate, completion rate, device usability, and outcome measures feasibility.

* Goal for recruitment: 100% of 30 subjects meeting all inclusion criteria can be recruited over the 36 week pilot recruitment phase.
* Completion and compliance: 90% of subjects will complete the study, 90% of sessions within each subject will be completed, and for completing subjects, 100% of measures will be completed.
* Useability: all therapists and subjects must rate useability as good or better.
* Success of blind: subject accuracy at guessing group membership must be at or near 50%.

ELIGIBILITY:
Inclusion Criteria:

1. Veteran or Servicemember
2. 18 to 50 years old
3. Sustained one or more mild traumatic brain injury (mTBI)s
4. Demonstration of balance deficits on the Sensory Organization Test (a composite score of 75 or less (1/3 sample) and 72 or less (2/3 sample))
5. Available for the duration of the study

Exclusion Criteria:

1. History of traumatic brain injury (TBI) of any severity other than mild TBI
2. Presence of active substance abuse condition
3. Any condition for which posturography is contraindicated (e.g. leg amputation or fracture)
4. Diagnosed neurological disorder with balance sequelae, other than TBI (e.g. Parkinson's disease, incomplete spinal cord injury, or Multiple Sclerosis)
5. Orthostatic hypotension as defined by:

   1. A systolic blood pressure decrease (from supine to sitting) of at least 20 mmHg
   2. A diastolic blood pressure decrease of at least 10 mmHg, or
   3. A pulse increase of 30 beats or more per minute with associated signs or symptoms of cerebral hypoperfusion
6. An implanted medical device
7. Pregnancy
8. Oral infection
9. Known transmissible disease (HIV, hepatitis, influenza, TB)
10. Exam signs of serious disorder other than mTBI as defined by facial asymmetry, hoarseness and dysarthria (e.g. tumor, stroke).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 36 weeks
  Number and percentage of subjects recruited over the 36 week pilot recruitment phase
Completion and compliance rates | Up to 12 weeks
  Number and percentage of subjects who complete the study
Usability rating | 12 weeks
  Number and percentage of subjects and therapists who rated usability as good or better.
Success of blinding | 12 weeks
  Number and percentage of subjects who accurately guess group membership
Change in Sensory Organization Test (SOT) | 12 weeks
  Comparison of the SOT score between the treatment group and sham group at the intermediate follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: David X Cifu, MD, Principal Investigator — VA Department of Physical Medicine and Rehabilitation; William C Walker, MD, Principal Investigator — Virginia Commonwealth University (VCU)
Locations (2):
- United States (2):
  - McGuire Veterans Affairs Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia